CLINICAL TRIAL: NCT05794087
Title: Activated Macrophages and Ozone Toxicity II
Brief Title: The Role of Macrophage Activation in Lung Injury Following Ozone Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Howard M. Kipen, MD, MPH, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro2022002024; R01ES004738 (NIH)
Record Dates: First submitted 2023-02-10; First posted 2023-03-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Air Pollution
Keywords: Macrophage
MeSH Terms: interventions — Environment, Controlled; Ozone

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either clean air or ozone for the first exposure then crossed over to the alternate arm for the second exposure.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and laboratory personnel will not be informed of the type of exposure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clean Air, Then Ozone (Experimental): Subjects will be exposed to clean air for 3 hours at the first exposure visit and 0.2ppm ozone for 3 hours at the second exposure visit. The visits will be at least 2 weeks apart.
  Interventions: Other: Clean Air; Other: Ozone
- Ozone, Then Clean Air (Experimental): Subjects will be exposed to 0.2 ppm ozone for 3 hours at the first exposure visit and clean air for 3 hours at the second exposure visit. The visits will be at least 2 weeks apart.
  Interventions: Other: Clean Air; Other: Ozone

INTERVENTIONS:
Other: Clean Air — Subjects will be exposed to clean air for 3 hours.
Other: Ozone — Subjects will be exposed to 0.2 ppm ozone for 3 hours.

SUMMARY:
The purpose of the study is to better understand the mechanisms of lung injury from ozone exposure. Subjects will participate in two exposure sessions: filtered air and 0.2 ppm ozone. The exposure visits will be at least 2 weeks apart. Subjects will be asked to produce sputum through coughing after each exposure. The samples will be analyzed for macrophage activity.

DETAILED DESCRIPTION:
Subjects will be asked to come to the Rutgers EOHSI clinical center (Piscataway, NJ) for 5 study visits. A physical exam to determine eligibility will be done at the first study visit. If the subject is healthy and able to produce a sputum sample, he/she will then be scheduled for 2 3-hour exposure visits, at least 2 weeks apart. One exposure will be to clean air and the other exposure will be to 0.2 ppm ozone. During the exposures, subjects will be requested to ride an exercise bicycle intermittently (approximately every 15 minutes). A follow-up visit for sputum collection will be scheduled either 24, 48, or 72 hours after each exposure visit. Blood and exhaled breath samples will also be collected at each visit.

ELIGIBILITY:
Exclusion Criteria:

* Cardiovascular disease
* Respiratory disease
* Recent (within 4 weeks) respiratory or COVID-19 symptoms
* Diabetes
* Pregnancy
* HIV Infection
* History of smoking within the past 5 years.
* Orthopedic or rheumatologic conditions which would interfere with cycle use
* Inability to produce a sputum plug at screening
* Daily use of antioxidant supplements, excluding those in a multivitamin. These supplements include Vitamin C or E, selenium, beta-carotene, lycopene, lutein, zeaxanthin and ginkgo biloba. Supplements taken less frequently but at least once a week will be reviewed by the principal investigator for eligibility determination.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic activity of inflammatory cells in induced sputum | Within 3 days of exposure
  The metabolic activity of inflammatory cells in sputum will be assessed by the measurement of ATP production. The measurement will be made on an Agilent Seahorse using a Mitoplate Assay.

CONTACTS AND LOCATIONS:
Overall Officials: Howard M Kipen, MD, Principal Investigator — Rutgers School of Public Health
Locations (1):
- Rutgers - EOHSI, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No